CLINICAL TRIAL: NCT01857882
Title: Breast Reconstruction Decision Workshop Pilot RCT (Randomized Controlled Trial)
Brief Title: Decision Support Workshop for Breast Reconstruction
Acronym: DSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-1027-CE
Record Dates: First submitted 2013-05-06; First posted 2013-05-20 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast reconstruction; shared decision making; decision support intervention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Support Workshop (Experimental): The decision support workshop will be 2 hours in duration on the morning of the consultation and will be facilitated by a dedicated social worker from psycho-oncology.
  Interventions: Other: Decision Support Workshop
- Standard Care (No Intervention): Routine pre-consultation education

INTERVENTIONS:
Other: Decision Support Workshop — Incorporates the key components of shared decision-making and decision support with the philosophy of delivering supportive care to cancer patients.
  * Surgeon (30 mins): treatment options for breast reconstruction with indications/ contraindications, advantages / disadvantages, expected post-operative course, aesthetic result and complications with probabilities
  * Registered nurse (30 mins): preparing for surgery, postoperative recovery and how to navigate the health care system
  * Social worker (30 mins): values clarification exercise
  * Breast reconstruction patient volunteer (30 mins) questions and answers about her personal experience
  Arms: Decision Support Workshop

SUMMARY:
The purpose of this study is to determine the effectiveness of a pre-consultation decision support workshop for breast reconstruction after breast cancer, in facilitating the decision-making process, compared to routine pre-surgical education.

DETAILED DESCRIPTION:
Postmastectomy breast reconstruction is becoming increasingly utilized in breast cancer patients to provide surgical restoration of the breast mounds. The breast reconstruction discussions can be highly complex, as there are many different techniques, timing, and complications that are unique to each procedure. However ¼ of women report being dissatisfied with some component of their cancer or reconstructive care. Failure of the physician to provide adequate information about treatment options is the most frequent source of cancer patient dissatisfaction and breast reconstruction patients have expressed a need for further information regarding the complex decision to pursue breast reconstruction. In such scenarios of complex medical decision-making, decision support techniques may be an effective solution to information provision and shared decision-making. As a result, the investigators developed a pre-consultation educational group intervention delivered in a group setting for women considering breast reconstruction, with the aims to fill an existing information-gap, promote high-quality decision-making and enhance decision self-efficacy and other decision measures. This pilot study will be the first step in the evaluation of the educational group intervention and the results will be used to determine the feasibility and inform the optimal design for a definitive randomized controlled trial. This study will first examine the feasibility and acceptability of the intervention through implementation in a pilot, mixed-methods, 1:1 allocation parallel-arm randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient age: 18 - 79 years at the time of consultation
* In situ or invasive biopsy confirmed breast adenocarcinoma
* Considered for immediate or delayed breast reconstruction
* First consultation for breast reconstruction

Exclusion Criteria:

* Chest wall or atypical breast malignancy (ex: angiosarcoma) or inflammatory adenocarcinoma of the breast
* Completion any phase of reconstruction, or for revision reconstruction
* Patient cannot read or write in English.
* Cognitive impairment or uncontrolled psychiatric diagnosis

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toni Zhong, MD, MHS, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Causarano N, Platt J, Baxter NN, Bagher S, Jones JM, Metcalfe KA, Hofer SO, O'Neill AC, Cheng T, Starenkyj E, Zhong T. Pre-consultation educational group intervention to improve shared decision-making for postmastectomy breast reconstruction: a pilot randomized controlled trial. Support Care Cancer. 2015 May;23(5):1365-75. doi: 10.1007/s00520-014-2479-6. Epub 2014 Oct 29. PMID 25351455
- [Derived] Platt J, Baxter N, Jones J, Metcalfe K, Causarano N, Hofer SO, O'Neill A, Cheng T, Starenkyj E, Zhong T. Pre-consultation educational group intervention to improve shared decision-making in postmastectomy breast reconstruction: study protocol for a pilot randomized controlled trial. Trials. 2013 Jul 6;14:199. doi: 10.1186/1745-6215-14-199. PMID 23829442
- See also: E-publication link — http://rd.springer.com/article/10.1007%2Fs00520-014-2479-6

RESULTS

PARTICIPANT FLOW:
Groups:
- Decision Support Workshop: The decision support workshop will be 2 hours in duration on the morning of the consultation and will be facilitated by a dedicated social worker from psycho-oncology.
  Decision Support Workshop: Incorporates the key components of shared decision-making and decision support with the philosophy of delivering supportive care to cancer patients.
  * Surgeon (30 mins): treatment options for breast reconstruction with indications/ contraindications, advantages / disadvantages, expected post-operative course, aesthetic result and complications with probabilities
  * Registered nurse (30 mins): preparing for surgery, postoperative recovery and how to navigate the health care system
  * Social worker (30 mins): values clarification exercise
  * Breast reconstruction patient volunteer (30 mins) questions and answers about her personal experience
Period: Overall Study
Arm/Group | Decision Support Workshop | Standard Care
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients reported baseline clinical characteristics. One patient in each arm did not have evaluable decisional self-efficacy and conflict scores post-treatment, so their baseline scores were not included in the analysis of these variables. Therefore, for these measures at baseline, n=19 in the standard care arm and n=20 in the workshop arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Support Workshop | Standard Care | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (5.5) | 51.5 (9.1) | 51.2 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 21 | 20 | 41
Decisional conflict Scale [Mean (Standard Deviation); unit: units on a scale] — Decisional conflict at baseline. Standard Care n=19, Decision Support Workshop n=20.
  The decisional conflict scale measures personal perceptions of uncertainty in choosing options. It is a 16-item 5-response instrument that reports a total score from 0 - 100 with higher scores indicating more conflict (items are summed, divided by 16 and multiplied by 25).
  units on a scale | 56.8 (18.0) | 41.3 (17.1) | 49.3 (19.0)

OUTCOME MEASURES:

1. Primary Outcome: Decision Self-efficacy Scale
Description: Decision self-efficacy (DSE) scale is a prospectively designed instrument to evaluate patient self-confidence in decision-making, including shared decision-making. It has been validated among women facing treatment decisions for osteoporosis and used in cancer patients. Psychometric evaluation has shown high levels of internal consistency (Cronbach alpha 0.90). Decision self-efficacy is correlated with decision conflict subscales of feeling informed (r = 0.47) and supported (r = 0.45). This instrument has never been tested in the breast cancer or breast reconstruction population.
  The total score is calculated by summing the 11 items, dividing by 11 and multiplying by 25. Scores range from 0 (extremely low self-efficacy) to 100 (extremely high self-efficacy).
  The mean and standard deviation (SD) were calculated at baseline and after the initial consultation. Change in score was defined as the difference in total score between baseline and after consultation.
Time Frame: Change from baseline decision self-efficacy at 1 week after surgical consultation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Support Workshop | Standard Care
Number analyzed (Participants) | 20 | 19
units on a scale | 5.7 (12.8) | 5.1 (9.8)

2. Secondary Outcome: Decision Conflict Scale
Description: Decision conflict scale measures personal perceptions of uncertainty in choosing options and has been demonstrated to be valid and responsive to change. The decisional conflict scale is a 16-item 5-response instrument that reports a score from 0 - 100 with higher scores indicating more conflict (items are summed, divided by 16 and multiplied by 25).
Time Frame: Change from baseline decision conflict at 1 week after surgical consultation
Reporting Status: Not Posted

3. Secondary Outcome: Decision Preference and Decision Choice
Description: Decision Preference and Decision Choice has been used as a primary and secondary outcome in studies of decision support interventions in cancer patients. It demonstrates good test-retest reliability (test-retest coefficient > 0.90) and is sensitive to change when measured before and after an intervention.
Time Frame: baseline
Reporting Status: Not Posted

4. Secondary Outcome: Patient Involvement in Care Scale (PICS)
Description: PICS is a measure of patient perception of involvement with her care, and has seven 5-point Likert scale items that assess the extent to which the patient asked questions, offered opinions, and expressed concerns when meeting with the surgeon.
Time Frame: T1 (1 week after surgical consultation)
Reporting Status: Not Posted

5. Secondary Outcome: Satisfaction With Information (Sub-scale of BREAST-Q)
Description: The BREAST-Q is a procedure-specific and validated PRO that measures Hr-QOL and patient satisfaction with breast reconstruction. The "Satisfaction with Information" Subscale specifically measures patient satisfaction with the preoperative information and care provided by the plastic surgeon and other members of the medical team. There are 15 items that use a four-level Likert scale response format, the score is transformed on a scale of 0 to 100 with higher scores indicating greater satisfaction.
Time Frame: T1 (1 week after surgical consultation)
Reporting Status: Not Posted

6. Secondary Outcome: Qualitative Interview Assessment
Description: A subgroup of participants allocated to both the experimental and usual care groups will be asked to participate in a brief qualitative telephone interview. Purposeful sampling will be used to recruit 5 patients from each group to achieve data saturation and variability. Telephone interviews will be conducted by a social worker trained in qualitative methods. All participants randomized to the workshop will additionally be asked to complete a written survey for evaluation of the intervention immediately after participation in the workshop.
Time Frame: Within three months after initial consultation
Reporting Status: Not Posted

7. Secondary Outcome: Uptake Rate of Breast Reconstruction-Service Outcome
Description: The uptake rate of breast reconstruction (if patients chose breast reconstruction or no reconstruction)
Time Frame: Six months after initial consultation
Reporting Status: Not Posted

8. Secondary Outcome: Length of Consultation-service Outcome
Description: The length of the initial consultation with the plastic surgeon, measured in minutes. Consultations are expected to be between 20-60 mins.
Time Frame: Duration of initial consultation
Reporting Status: Not Posted

9. Secondary Outcome: Number of Consultations-service Outcomes
Description: The number of consultations with the plastic surgeon until the patient has made a reconstruction choice (defined as signing a surgical consent form) will be recorded. Patients can spend months considering their choices, so it is appropriate to follow them for a period of at least six months after their initial consultation.
Time Frame: Six months after initial consultation
Reporting Status: Not Posted

10. Secondary Outcome: Breast Reconstruction Knowledge Test
Description: This breast reconstruction knowledge test is a 12-item 3-response questionnaire that records the score on a continuous integer scale, and measured patient's knowledge regarding breast reconstruction.
Time Frame: Change in baseline breast reconstruction knowledge at 1 week after initial consultation
Reporting Status: Not Posted

11. Secondary Outcome: Medical Outcomes Study Social Support Survey
Description: Medical Outcomes Study Social Support Survey has a series of 18 questions that measure 4 domains of social support (emotional, tangible, affectionate, and social interactions). Responses range from 1 (none of the time) to 5 (all the time). The items in each domain were summed and then transformed to yield scores ranging from 0 to 100. Higher scores indicate more support.
Time Frame: baseline
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Recruitment Rate-feasibility Outcome
Description: As this is a pilot study, the feasibility of conducting the study is highly important. The recruitment rate of participants will be measured, during the recruiting period which is expected to be on average two months.
Time Frame: Duration of recruiting, expected on average two months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Retention After Randomized Treatment Assignment (Workshop and Consultation Attendance)-Feasibility Outcome
Description: The number of participants who completed their assigned treatment (workshop and consultation vs. consultation alone) will be recorded. This will be recorded directly after each day the treatment is delivered.
Time Frame: Duration of treatment-8 hours on day of treatment
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Completion of Primary Outcome Measure-feasibility Outcome
Description: Patients are to complete the primary outcome one week after initial consultation. However, it is expected that some patients may take longer to complete this intervention (on average 1 month after consultation), and will require reminder telephone calls.
Time Frame: 1 week after initial consultation
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse events were not assessed. Patients were not at risk for adverse events from this intervention ( 2 hour group workshop), as it was not medically invasive.
Arm/Group | Decision Support Workshop | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No